CLINICAL TRIAL: NCT06552390
Title: Cardiac Rehabilitation for Inpatient Heart Transplant (HRN4HTx)
Acronym: HRN4HTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Bragança (Other)
Collaborators: Unidade Local de Saúde de Coimbra (Unknown); Universidade do Porto (Other)
Responsible Party: Principal Investigator, André Filipe Morais Pinto Novo, Coordinator Professor, Instituto Politécnico de Bragança
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRN4HTx_1.0
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Heart Transplantation
Keywords: Cardiac Rehabilitation; Rehabilitation; Self Care
MeSH Terms: interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group - HRN4HTx (Experimental): Cardiac rehabilitation as previously described.
  Interventions: Procedure: Cardiac Rehabilitation

INTERVENTIONS:
Procedure: Cardiac Rehabilitation — HRN4HTx is a phase 1 rehabilitation intervention protocol for post-heart transplant focused on the physical exercise component, and an educational plan regarding risk factors and safety criteria. The intervention protocol and its assessments are implemented by the team's rehabilitation nurses, always safeguarding the protective isolation required for these patients. The physical training protocol is divided into five stages of progressive levels of intervention. The protocol was defined following FITT parameters, international recommendations, and an integrated teaching program aimed at the therapeutic regimen exercise area. The frequency of intervention sessions is 7 days a week, twice a day (average of 13 sessions per week) throughout the hospitalization.
  The intensity was defined according to Borg's modified scale of subjective perception of exertion (SPE), which must be maintained at less than 5.

SUMMARY:
To evaluate the safety and efficacy of the phase 1 cardiac rehabilitation protocol(HRN4HTx) in heart transplant patients, focusing on self-care capacity and functionalrecovery.

DETAILED DESCRIPTION:
Type of study: Descriptive and Interventional Study

- Location: Centro Hospitalar e Universitário de Coimbra, Cardiothoracic Surgery Unit

Study Population:

* Inclusion Criteria: Heart transplant patients, over 18 years of age, capable of providing informed consent.
* Exclusion Criteria: Rejection 2R, inability to understand due to cognitive impairment, external ventricular assistance, infectious processes with hemodynamic changes.

Intervention:

The HRN4HTx protocol was implemented during hospitalization, divided into five progressive stages according to FITT parameters and international recommendations. Interventions included respiratory exercises, calisthenics exercises, balance training, resistance exercises for upper and lower limbs, and walking.

Adverse Event Monitoring:

Adverse events (AEs) and serious adverse events (SAEs) were monitored according to Good Clinical Practices. Examples of monitored events include arrhythmias and significant changes in blood pressure.

Outcomes Measured:

* Self-Care Capacity: Barthel Index measured at admission and discharge.
* Functional Capacity: 6-minute walk test (6MWT) conducted at discharge.
* Knowledge of Risk Factors: Evaluation of knowledge regarding alarm signs and cardiovascular risk factors at discharge.

Ethical Approval:

This study was approved by the Ethics Committee of the Centro Hospitalar e Universitáriode Coimbra (Protocol No. OBS.SF.111/2021). All participants provided written informed consent prior to participation.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant patients, over 18 years of age, capable of providing informedconsent.

Exclusion Criteria:

* Rejection 2R
* Inability to understand due to cognitive impairment
* External ventricular assistance
* Infectious processes with hemodynamic changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Functional Capacity - Evaluation of the 6-minute walk test (6MWT) | At the date of discharge (mean days of hospitalization of 15 until a maximum of days 21)
  6-minute walk test (6MWT), higher value means better outcome (no maximum value)
Self-Care Capacity - Evaluation of the Barthel Index | At the date of admission and at the date of discharge (mean days of hospitalization of 15 until a maximum of 21 days)
  Barthel Index, from 0 to 100, higher scores means better outcome
Knowledge of Risk Factors - Evaluation of knowledge regarding alarm signs and cardiovascular risk factors | At the date of discharge (mean days of hospitalization of 15 until a maximum of 21 days)
  Knowledge regarding alarm signs and cardiovascular risk factors, from 0 to 100%, higher value means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: André Novo, PhD., Study Director — Instituto Politécnico de Bragança
Locations (1):
- Unidade Local de Saúde de Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loureiro M, Parola V, Duarte J, Oliveira I, Antunes M, Coutinho G, Martins MM, Novo A. Cardiac Rehabilitation to Inpatient Heart Transplant-HRN4HTx Intervention Protocol. Nurs Rep. 2024 Aug 23;14(3):2084-2094. doi: 10.3390/nursrep14030155. PMID 39311164